CLINICAL TRIAL: NCT04423276
Title: Efficiency of Donepezil in Elderly Patients Undergoing Orthopedic Surgery Due to Underlying Postoperative Cognitive Dysfunction, a Multicenter Randomized Controlled Trial
Brief Title: Efficiency of Donepezil in Elderly Patients for Prevention of POCD Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other); Tenth People's Hospital of Tongji Univeristy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DNPQ20200523
Record Dates: First submitted 2020-06-06; First posted 2020-06-09 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Total Knee Arthroplasty; Fracture of Head of Femur Articular Displaced; Protrusion of Intervertebral Disc
MeSH Terms: interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Drug: Placebo
- Donepezil (Experimental)
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Donepezil a cholinesterase inhibitor, 5mg(1 pill)/ day for 7 days Po, was administrated from the day before surgery.
  Arms: Donepezil
Drug: Placebo — Placebo, 1 pill/ day for 7 days Po, was administrated from the day before surgery.
  Arms: Control

SUMMARY:
Postoperative cognitive dysfunction (POCD) occurs mainly in aged patients. POCD may increase the mortality and morbidity. However, the mechanism of POCD is not clear yet and no effective therapy method was proved. According to our previous study, the central cholinergic system impaired by the anesthesia and surgery play a very important role in the POCD and donepezil an acetylcholinesterase inhibitor can prevent the POCD after isoflurane anesthesia in aged mice. Donepezil is a commercial medicine used for the Alzheimer Disease, which is tolerable and has minimal adverse events. In present study a multi-center randomized case control study was conducted and we hypothesized that donepezil attenuate the POCD.

ELIGIBILITY:
Inclusion Criteria:

1. Elder than 60 years old
2. Speak Chinese Mandarin
3. Scheduled to undergo hip or knee replacement surgery and lumbar spine surgery
4. The operation time is more than 2 hours.
5. Signed the informed consent
6. American Society of Anesthesiologists (ASA) classification I-II

Exclusion Criteria:

1. Existing cerebral disease, or have a history of neurological and psychiatric diseases including Alzheimer Disease, stroke, epilepsy and psychosis
2. Existing cognitive impairment as evidenced by Mini-Mental State Examination scores below 24
3. Several audition or vision disorder
4. Patients with tumors or infections
5. Unwillingness to comply with the protocol or procedures
6. Can not communicate normally in Mandarin Chinese
7. Existing bradycardiac arrhythmia (Heart rate <60 bpm for any reasons)
8. Existing gastrointestinal ulcer
9. Existing urinary incontinence
10. Existing asthma or chronic obstructive pulmonary disease
11. Postoperative admission to ICU
12. Allergic to donepezil

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-06-14 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of POCD after the surgery. | up to 7 days

SECONDARY OUTCOMES:
The incidence of postoperative delirium after surgery. | 1 to 7 days after surgery
POCD incidence one month, six months and one year after surgery. | one month, six months and one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Principal Investigator — Department of Anesthesiology Renji Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhu H, Cong L, Chen Y, Chen S, Chen L, Huang Z, Zhou J, Xiao J, Huang Y, Su D. Efficiency of donepezil in elderly patients undergoing orthopaedic surgery due to underlying post-operative cognitive dysfunction: study protocol for a multicentre randomised controlled trial. Trials. 2021 Oct 9;22(1):688. doi: 10.1186/s13063-021-05648-0. PMID 34627332